CLINICAL TRIAL: NCT06840184
Title: Culturally Adapted Cognitive Behavioral Therapy Based Self Help Intervention for Mental Health of Caregivers of Individuals With Substance Use: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatima Jinnah Women University (Other)
Responsible Party: Principal Investigator, Jawairia Zia, Principal Investigator, Fatima Jinnah Women University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: FJWU/EC/2025/103
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Psychological Stress; Quality of Life (QOL); Mental Health
Keywords: Khushi Aur Khatoon; CBT Self Help intervention
MeSH Terms: conditions — Stress, Psychological; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group which received intervention (Experimental): The experimental group was provided with CBT Self- help Intervention (Khushi aur Khatoon), a 4-6 weeks program for improvement of emotional resilience and mental well- being.
  Interventions: Behavioral: Cognitive Behavioral Therapy based Intervention
- Control Group (Active Comparator): No intervention was provided to the control group, except for a few members who requested for the therapy, that too after the post assessment.
  Interventions: Other: No intervention

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy based Intervention — Session 1: Introduction of CBT, Relationship between events, thoughts and behavior.
  Session 2: Psychoeducation about the vicious circle of inactivity and depression, Ladder technique for task management.
  Session 3: Problem solving techniques and discussion about them, Decision making techniques through "Advantages/ Disadvantages" chart.
  Session 4: Identifying positive and negative emotions, Cognitive errors were explained.
  Session 5: Identifying negative thoughts through Socratic questioning, Finding evidence for and against the thoughts, Challenging negative thought, Cracking firm irrational beliefs.
  Session 6: Cognitive restructuring techniques, Finding alternative thoughts.
  Arms: Experimental Group which received intervention
Other: No intervention — No intervention was provided to the control group, except for a few members who requested for the therapy, that too after the post assessment.
  Arms: Control Group

SUMMARY:
The primary purpose of this study is to investigate whether Cognitive Behavioral Therapy based Self- Help Intervention can significantly reduce emotional problems as well as improve the mental well being and quality of life among the caregivers of individuals with substance use. The study aims to contribute to the existing literature by providing evidence on the efficacy of the above mentioned therapy. This can be helpful in improving clinical practices and treatment outcomes.

DETAILED DESCRIPTION:
The current quantitative study comprises of two phases. Pilot study for translation and validation of scales were done as a preliminary step. The first phase was a cross-sectional survey to screen out potential caregivers of substance users, with depression, anxiety and stress, higher than the normal level. A randomized controlled trial (RCT) was done in the second phase, where caregivers of substance users who had higher level of psychological distress, were categorized into two groups; control group and intervention group through randomization. Cognitive Behavioral Therapy based intervention (Self- Help Manuel named, "Khushi aur Khatoon") was provided to the intervention group in 4-6 individual and face to face sessions. Control group did not receive therapy ( on request of some of the members of control group, therapy was provided after the completion of the study). Pre and post- assessment of the study variables were done for both control and intervention groups. Difference between pre and post assessment was compared to investigate the effectiveness of Cognitive Behavioral Therapy based intervention ("Khushi aur Khatoon") among caregivers of substance users.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 and above.
* Those who will have burden and distress above the normal levels on respective scales during baseline assessment.
* Capable of providing written informed consent.
* Residing within the catchment areas of the participating rehabilitation center.

Exclusion Criteria:

* Individuals unable to provide consent due to severe mental or physical illness.
* Individuals not capable of reading and comprehending Urdu versions of the intervention manual and scales.
* Unlikely to be accessible for outcome assessments due to temporary residence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
DASS- 21 (Urdu) | 3 months
  This scale has 21- Items comprising of 3 subscales, designed to assess emotional states related to depression, anxiety, and stress (7 items each). Higher scores on the scale indicate higher levels of psychological distress and low scores indicate low psychological distress.
Quality of Life Questionnaire (Urdu) | 3 months
  It is a 15-item instrument consisting of four domains: physical health, psychological health, social relationships, and environmental health; it also contains QOL and general health items. Higher score on QOLQ represents higher quality of life, whereas low scores depict low quality of life.
Caregivers' Burden Questionnaire (Urdu) | 3 months
  This scale measures two aspects of burden (objective and subjective) comprising of 6 items each. This scale encompasses financial burden, disruption of routine family activities, family leisure, family interactions, and effect on physical and mental health of caregivers. Higher score on Caregivers' Burden Questionnaire represents higher level of burden caregivers, whereas low scores depict low caregivers' burden
Warwick- Edinburgh Mental Well- Being Scale (Urdu) | 3 months
  The 14- items scale covers subjective well- being and psychological functioning. Higher score on the scale represents higher level of mental well- being, whereas low scores depict low mental well- being.

SECONDARY OUTCOMES:
Role Burden Scale (Urdu) | 3 months
  It measures the psychological as well as physical burden on a person due to performing multiple roles in their daily routine. Only "Item # 1" has to be scored in reverse manner. Higher score on Role Burden Scale represents higher burden on the participant due to holding multiple roles, whereas low scores depict low role burden

CONTACTS AND LOCATIONS:
Overall Officials: Jawairia Zia, M Phil, Principal Investigator — Fatima Jinnah Women University
Locations (1):
- Islah drug Rehabilitation Center, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Due to ethical concerns, data will not be shared. All research findings will be published in aggregate form maintaining anonymity of the participants.

REFERENCES:
- [Background] Amin R, Iqbal A, Naeem F, Irfan M. Effectiveness of a culturally adapted cognitive behavioural therapy-based guided self-help (CACBT-GSH) intervention to reduce social anxiety and enhance self-esteem in adolescents: a randomized controlled trial from Pakistan. Behav Cogn Psychother. 2020 Sep;48(5):503-514. doi: 10.1017/S1352465820000284. Epub 2020 May 26. PMID 32450939
- See also: Effectiveness of a culturally adapted cognitive behavioural therapy-based guided self-help (CACBT-GSH) intervention to reduce social anxiety and enhance self-esteem in adolescents: a randomized controlled trial from Pakistan. — https://pubmed.ncbi.nlm.nih.gov/32450939/